CLINICAL TRIAL: NCT02092038
Title: Phase I Pilot Study of Preoperative Chemoradiation for Glioblastoma
Brief Title: Preoperative Chemoradiation for Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tampa General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGH0001
Record Dates: First submitted 2014-03-11; First posted 2014-03-19 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Glioblastoma
Keywords: glioblastoma; temozolomide; radiation therapy; radiotherapy; surgery; pre-operative; neoadjuvant
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Craniotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preoperative chemoradiation (Experimental): Stereotactic biopsy of brain tumor, then partial brain irradiation and temozolomide, followed by craniotomy and tumor resection, followed by temozolomide
  Interventions: Drug: Temozolomide; Radiation: partial brain irradiation; Procedure: stereotactic biopsy of brain tumor; Procedure: craniotomy and tumor resection

INTERVENTIONS:
Drug: Temozolomide — Neoadjuvant treatment with concurrent temozolomide and radiation therapy, followed by surgery and then further temozolomide.
  Other Names: Temodar
Radiation: partial brain irradiation — Neoadjuvant treatment with concurrent temozolomide and radiation therapy, followed by surgery and then further temozolomide.
Procedure: stereotactic biopsy of brain tumor — will be assessed for tumor type and tumor markers
Procedure: craniotomy and tumor resection — maximal safe resection

SUMMARY:
Trial to determine the safety of neoadjuvant treatment with concurrent temozolomide and radiation therapy, followed by surgery and then further temozolomide.

DETAILED DESCRIPTION:
Prior to any definitive treatment and after enrollment, the patient will undergo stereotactic biopsy of the lesion to confirm the histology of the lesion and to determine methylated methylguanine methyltransferase (MGMT) status. Standard image-guided stereotactic technique will be used. Patients will be treated with conformal radiation therapy. Temozolomide will be given from the day prior to radiation therapy through the last day of radiation therapy. 4-6 weeks after radiation therapy the patient will undergo craniotomy and maximal safe resection. Temozolomide will continue beginning 4 weeks after surgery.

Imaging:

MRI within 2 weeks prior to the start of the protocol. MRI at 4 weeks after chemoradiation therapy and prior to surgery. MRI within 48 hours after surgery.

MRI after every 2 cycles of chemotherapy and then every 2 months until progression, up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* MRI lesions of the brain that have a high probability of being glioblastoma in a potentially resectable location in the brain (the primary study population)
* WHO performance status 0-2 (to allow comparison to historical controls)
* Adequate hematological parameters: (for safety because of neutropenia from the temozolomide)
* Consent can be obtained from the patient, and if the patient cannot give consent then from the medical power of attorney and if one is not assigned, then the nearest relative (required to obtain consent)
* Able to have MRI scans (secondary endpoint is MRI scan characteristics)
* Willing to have radiation treatment at a participating center (homogeneity of treatment parameters)
* Ages 18-80

Exclusion Criteria:

* Unresectable tumor
* Absolute neutrophil count (ANC) less than 1,200/μL
* Hemoglobin less than 9.0g/dL
* Platelet count less than 100,000/μL

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
toxicity of treatment per Common Toxicity Criteria for Adverse Effects V3.0 | up to up to 16 weeks
  comparison of toxicity related to experimental treatment to historical local controls

SECONDARY OUTCOMES:
Feasibility of measurement of O(6)-Methylguanine-DNA methyltransferase (MGMT) activity on stereotactic samples | at enrollment
  determination of the feasibility of using standard MGMT activity measurement techniques on stereotactic specimens and comparison of the results with the results from the full resection.
progression free survival | up to 12 months
overall survival | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Berk, MD, PhD, Principal Investigator — Tampa General Hospital
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States